CLINICAL TRIAL: NCT04376684
Title: A Randomized, Double-blind, Placebo-controlled, Study Evaluating the Efficacy and Safety of Otilimab IV in Patients With Severe Pulmonary COVID-19 Related Disease
Brief Title: Investigating Otilimab in Patients With Severe Pulmonary COVID-19 Related Disease
Acronym: OSCAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 214094
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Severe Acute Respiratory Syndrome
Keywords: COVID-19; Otilimab; Ordinal scale; Coronavirus; GSK3196165
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Coronavirus Infections | interventions — Otilimab; Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either a blinded IV infusion of otilimab or placebo, in addition to standard of care.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Participants receiving otilimab (Experimental): Participants (age >=18 years and <=79 years) will receive a single dose of otilimab administered as an IV infusion in addition to standard of care in Part 1.
  Interventions: Biological: Otilimab; Drug: Standard of care
- Part 1: Participants receiving placebo 1 (Placebo Comparator): Participants (age >=18 years and <=79 years) will receive a single dose of matching placebo administered as an IV infusion in addition to standard of care in Part 1.
  Interventions: Biological: Placebo 1; Drug: Standard of care
- Part 2: Participants receiving otilimab (Experimental): Participants (age 70 years or above) will receive a single dose of otilimab administered as an IV infusion in addition to standard of care in Part 2.
  Interventions: Biological: Otilimab; Drug: Standard of care
- Part 2: Participants receiving placebo 2 (Placebo Comparator): Participants (age 70 years or above) will receive a single dose of matching placebo administered as an IV infusion in addition to standard of care in Part 2.
  Interventions: Biological: Placebo 2; Drug: Standard of care

INTERVENTIONS:
Biological: Otilimab — Otilimab will be administered once via IV route.
  Arms: Part 1: Participants receiving otilimab; Part 2: Participants receiving otilimab
Biological: Placebo 1 — Placebo 1 will consist of sterile 0.9 percent (%) sodium chloride solution administered once via IV route.
  Arms: Part 1: Participants receiving placebo 1
Biological: Placebo 2 — Placebo 2 will consist of sterile 5% dextrose or 5% glucose solution administered once via IV route.
  Arms: Part 2: Participants receiving placebo 2
Drug: Standard of care — All participants will receive standard of care as per institutional protocol.

SUMMARY:
OSCAR (Otilimab in Severe COVID-19 Related Disease) is a multi-center, double-blind, randomized, placebo-controlled trial to assess the efficacy and safety of otilimab for the treatment of severe pulmonary COVID-19 related disease. The study is being conducted in 2 parts (Part 1 and Part 2). Otilimab is a human monoclonal anti-granulocyte macrophage colony stimulating factor (GM-CSF) antibody that has not previously been tested in participants with severe pulmonary COVID-19 related disease in Part 1. The aim of this study is to evaluate the benefit-risk of a single infusion of otilimab in the treatment of hospitalized participants with severe COVID-19 related pulmonary disease with new onset hypoxia requiring significant oxygen support or requiring early invasive mechanical ventilation (less than or equal to [<=] 48 hours before dosing). Participants will be randomized to receive a single intravenous (IV) infusion of otilimab or placebo, in addition to standard of care.

ELIGIBILITY:
Inclusion criteria for Part 1:

* Participants aged >=18 years and <=79 years at the time of obtaining informed consent.
* Participants must:

  1. have positive severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) result (any validated test, for example. reverse transcription polymerase chain reaction [RT-PCR] [performed on an appropriate specimen; for example: respiratory tract sample])
  2. and be hospitalized due to diagnosis of pneumonia (chest X-ray or computerized tomography [CT] scan consistent with COVID-19)
  3. and be developing new onset of oxygenation impairment requiring any of the following:

     1. high-flow oxygen (>=15L/min)
     2. non-invasive ventilation (for example. CPAP, BIPAP)
     3. mechanical ventilation <=48 hours prior to dose
  4. and have increased biological markers of systemic inflammation (either C-reactive protein [CRP] >upper limit of normal [ULN] or serum ferritin >ULN).
* No gender restriction.
* Female participants must meet and agree to abide by the contraceptive criteria detailed in the protocol. Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* A female participant is eligible to participate if she is not pregnant or breastfeeding or if she is using highly effective contraceptive methods. Women of non-childbearing potential can also participate. A negative highly sensitive pregnancy test at hospital admission or before the first dose of study intervention.
* Capable of giving written informed consent.

Inclusion Criteria for Part 2:

* Participants aged 70 years or above at the time of obtaining informed consent.
* Participants must:

  1. have positive SARS-CoV-2 result (any validated test, for example. RT-PCR [performed on an appropriate specimen; for example. respiratory tract sample])
  2. and be hospitalized due to diagnosis of pneumonia (chest X-ray or CT scan consistent with COVID-19).
  3. and be developing new onset of oxygenation impairment requiring any of the following:

     1. high-flow oxygen (>=15L/min)
     2. non-invasive ventilation (for example. CPAP, BiPAP)
     3. mechanical ventilation <=48 hours prior to dose
  4. and have increased biological markers of systemic inflammation (either CRP >ULN or serum ferritin >ULN.
* No gender restriction.
* Capable of giving written informed consent.

Exclusion Criteria for Part 1:

* Progression to death is imminent and inevitable within the next 48 hours, irrespective of the provision of treatments, in the opinion of the investigator.
* Multiple organ failure according to the investigator's judgement or a Sequential Organ Failure assessment (SOFA score) >10 if in the ICU.
* Extracorporeal membrane oxygenation (ECMO) hemofiltration/dialysis or high-dose (>0.15 micrograms [mcg]/kilograms [kg]/min) noradrenaline (or equivalent) or more than one vasopressor.
* Current serious or uncontrolled medical condition (for example: significant pulmonary disease [such as severe chronic obstructive pulmonary disease (COPD) or pulmonary fibrosis], heart failure [New York Heart Association {NYHA} class III or higher], renal dysfunction, acute myocardial infarction or acute cerebrovascular accident within the last 3 months) or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study.
* Untreated systemic bacterial, fungal, viral, or other infection (other than SARS-CoV-2).
* Known active tuberculosis (TB), history of untreated or incompletely treated active or latent TB, suspected or known extrapulmonary TB.
* Known Human Immunodeficiency Virus (HIV) regardless of immunological status.
* Known hepatitis B surface antigen (HBsAg) and/or anti-hepatitis C virus (HCV) positive.
* Currently receiving radiotherapy, chemotherapy or immunotherapy for malignancy.
* Received monoclonal antibody therapy (for examplee. tocilizumab, sarilumab) within the past 3 months prior to randomization, including intravenous immunoglobulin, or planned to be received, during the study.
* Received immunosuppressant therapy including but not limited to cyclosporin, azathioprine, tacrolimus, mycophenolate, Janus Kinase (JAK) inhibitors (for examplee. baricitinib, tofacitinib, upadacitinib) within the last 3 months prior to randomization or planned to be received during the study.
* History of allergic reaction, including anaphylaxis to any previous treatment with an anti-GM-CSF therapy.
* Received COVID-19 convalescent plasma within 48 hours of randomization.
* Currently receiving chronic oral corticosteroids for a non-COVID-19 related condition in a dose higher than prednisone 10 milligrams (mg) or equivalent per day.
* Treatment with an investigational drug within 30 days of randomization.
* Participating in other drug clinical trials, including for COVID-19.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5 times ULN.
* Platelets <50,000/cubic millimeters (mm^3)
* Hemoglobin <=9 grams per deciliter (g/dL)
* Absolute neutrophil count (ANC) <1.5 times 10^9/L (neutropenia >= Grade 2)
* Estimated glomerular filtration rate (GFR) <=30 milliliters (mL)/min/1.73 meter square (/m^2).
* Pregnant or breastfeeding females.

Exclusion Criteria for Part 2:

* Progression to death is imminent and inevitable within the next 48 hours, irrespective of the provision of treatments, in the opinion of the investigator.
* Multiple organ failure according to the investigator's judgement or a SOFA score >10 if intubated in the ICU.
* ECMO hemofiltration/dialysis, or more than one inotrope/vasopressor of any class.
* Current serious or uncontrolled medical condition (for example. significant pulmonary disease [such as severe COPD or pulmonary fibrosis], heart failure [NYHA class III or higher], severe renal dysfunction, acute myocardial infarction or acute cerebrovascular accident within the last 3 months), severe dementia, severe disability, or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study.
* Untreated systemic bacterial, fungal, viral, or other infection (other than SARSCoV-2).
* Known active TB, history of untreated or incompletely treated active or latent TB, suspected or known extrapulmonary TB.
* Known HIV regardless of immunological status.
* Known HBsAg and/or anti-HCV positive (participants demonstrating a sustained virologic response (SVR) are not excluded from participation).
* Currently receiving radiotherapy, chemotherapy (hormone based therapies are permitted) or immunotherapy for malignancy.
* Received monoclonal antibody therapy (for example. tocilizumab, sarilumab) within the past 3 months prior to randomization, including intravenous immunoglobulin, or planned to be received during the study.
* Received immunosuppressant therapy including but not limited to cyclosporin, azathioprine, tacrolimus, mycophenolate, JAK inhibitors (for example. baricitinib, tofacitinib, upadacitinib), nintedanib, disease modifying antirheumatic drugs (DMARDs) (for example. methotrexate) within the last 3 months prior to randomization or planned to be received during the study.
* History of allergic reaction, including anaphylaxis to any previous treatment with an anti-GM-CSF therapy.
* Received COVID-19 convalescent plasma within 48 hours of randomization.
* Currently receiving chronic oral corticosteroids for a non-COVID-19 related condition at a dose higher than prednisone 10 mg or equivalent per day.
* Treatment with an investigational drug or substance within 30 days of randomization unless approved by the Medical Monitor.
* Participating in other drug clinical trials, including for COVID-19.
* AST or ALT >5 times ULN.
* Platelets <50,000/mm^3.
* Hemoglobin <=9 g/dL
* ANC <1.0 x 10^9/L (neutropenia >= Grade 3).
* Estimated GFR <=30 mL/min/1.73 m^2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1156 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (100):
- United States (21):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Winfield, Illinois
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Germantown, Maryland
  - GSK Investigational Site, Silver Spring, Maryland
  - GSK Investigational Site, Saint Louis Park, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Reno, Nevada
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Doylestown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (4):
  - GSK Investigational Site, Munro, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Yvoir
- Brazil (3):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São Paulo
- Canada (5):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Jérôme, Quebec
- GSK Investigational Site, Santiago, Chile
- GSK Investigational Site, Bogotá, Colombia
- France (11):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Argenteuil
  - GSK Investigational Site, La Roche-sur-Yon
  - GSK Investigational Site, La Tronche
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Melun
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Valenciennes
- India (7):
  - GSK Investigational Site, Aurangabad
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
- GSK Investigational Site, Napoli, Campania, Italy
- Japan (5):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- Mexico (4):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Mexico City, Mexico City
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México
- Netherlands (5):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
- GSK Investigational Site, Lima, Peru
- Poland (5):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Russia (10):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yekaterinburg
- South Africa (6):
  - GSK Investigational Site, Benoni, Gauteng
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Panorama
  - GSK Investigational Site, Tygerberg
  - GSK Investigational Site, Worcester
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Logroño
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, San Sebastián de Los Reyes/Madrid
- United Kingdom (3):
  - GSK Investigational Site, Manchester, Greater Manchester
  - GSK Investigational Site, Newcastle, Northumberland
  - GSK Investigational Site, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Background] Patel J, Bass D, Beishuizen A, Bocca Ruiz X, Boughanmi H, Cahn A, Colombo H, Criner GJ, Davy K, de-Miguel-Diez J, Doreski PA, Fernandes S, Francois B, Gupta A, Hanrott K, Hatlen T, Inman D, Isaacs JD, Jarvis E, Kostina N, Kropotina T, Lacherade JC, Lakshminarayanan D, Martinez-Ayala P, McEvoy C, Meziani F, Monchi M, Mukherjee S, Munoz-Bermudez R, Neisen J, O'Shea C, Plantefeve G, Schifano L, Schwab LE, Shahid Z, Shirano M, Smith JE, Sprinz E, Summers C, Terzi N, Tidswell MA, Trefilova Y, Williamson R, Wyncoll D, Layton M. A randomised trial of anti-GM-CSF otilimab in severe COVID-19 pneumonia (OSCAR). Eur Respir J. 2023 Feb 2;61(2):2101870. doi: 10.1183/13993003.01870-2021. Print 2023 Feb. PMID 36229048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-part study evaluating efficacy and safety of intravenously (IV) administered otilimab in participants with severe pulmonary Coronavirus Disease-2019 (COVID-19) related disease. Part 1 consisted of participants aged 18 to 79 years and Part 2 consisted of participants aged 70 years and older.
Pre-assignment Details: A total of 1156 (806 in Part 1 and 350 in Part 2) participants were enrolled in the study (Enrolled Population: All participants who entered the study).
Groups:
- Part 1: Placebo 1: Participants between the ages of greater than or equal to (>=)18 years and less than or equal to (<=)79 years received blinded 1-hour IV infusion of placebo (sterile 0.9 percent [%] weight by volume [w/v] sodium chloride solution) once along with standard of care.
- Part 1: Otilimab 90 mg: Participants between the ages of >=18 years and <=79 years received blinded otilimab 90 milligrams (mg) (solution in single-use vial diluted in sterile 0.9% w/v sodium chloride solution) once as 1-hour IV infusion along with standard of care.
- Part 2: Placebo 2: Participants aged 70 years or above received blinded 1-hour IV infusion of placebo (sterile 5% w/v dextrose solution) once along with standard of care.
- Part 2: Otilimab 90 mg: Participants aged 70 years or above received blinded otilimab 90 mg (solution in single-use vial diluted in sterile 5% dextrose solution) once as 1-hour IV infusion along with standard of care.
Period: Part 1 (Up to Day 60)
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Started | 403 | 403 | 0 | 0
Completed | 388 | 379 | 0 | 0
Not Completed | 15 | 24 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 8 | 0 | 0
Not completed — Protocol Violation | 2 | 3 | 0 | 0
Not completed — Physician Decision | 2 | 5 | 0 | 0
Not completed — Lost to Follow-up | 4 | 8 | 0 | 0
Period: Part 2 (Up to Day 60)
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Started | 0 | 0 | 175 | 175
Completed | 0 | 0 | 170 | 171
Not Completed | 0 | 0 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were presented for Enrolled Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg | Part 2: Placebo 2 | Part 2: Otilimab 90 mg | Total
Number analyzed (Participants) | 403 | 403 | 175 | 175 | 1156
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0
  Between 18 to 64 years | 249 | 250 | 0 | 0 | 499
  >=65 to 84 years | 154 | 153 | 168 | 168 | 643
  >=85 years | 0 | 0 | 7 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 101 | 75 | 73 | 377
  Male | 275 | 302 | 100 | 102 | 779
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 30 | 3 | 8 | 65
  Asian - Central/South Asian Heritage | 42 | 31 | 1 | 0 | 74
  Asian - East Asian Heritage | 4 | 4 | 0 | 0 | 8
  Asian - Japanese Heritage | 15 | 14 | 13 | 5 | 47
  Asian - South East Asian Heritage | 12 | 8 | 1 | 0 | 21
  Black or African American | 25 | 26 | 6 | 6 | 63
  White - Arabic/North African Heritage | 27 | 21 | 14 | 21 | 83
  White - White/Caucasian/European Heritage | 235 | 251 | 136 | 134 | 756
  Mixed Asian Race | 0 | 1 | 0 | 0 | 1
  Mixed White Race | 1 | 1 | 1 | 0 | 3
  Multiple | 7 | 7 | 0 | 0 | 14
  Unknown | 11 | 9 | 0 | 1 | 21

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants Alive and Free of Respiratory Failure at Day 28
Description: Participants were considered alive and free of respiratory failure if they were in category 1, 2, 3, or 4 from the GlaxoSmithKline (GSK) modified version ordinal scale adapted from World Health Organization (WHO) scale 2020. The 8-point scale was as follows: 1) Non-hospitalized, no limitation of activity; 2) Non-hospitalized,limitation of activity; 3) Hospitalized, no oxygen therapy; 4) Hospitalized, low-flow oxygen by mask or nasal prongs; 5) Hospitalized, highflow oxygen (greater than or equal to [>=]15 liters per minute [L/min]), continuous positive airway pressure (CPAP), bilevel positive airway pressure (BIPAP), non-invasive ventilation; 6) Hospitalized, intubation and mechanical ventilation; 7) Hospitalized, mechanical ventilation plus additional organ support; 8) Death. Higher scale indicates higher intensity of respiratory failure. Percentage values are rounded off.
Time Frame: At Day 28
Population: Modified intent to treat (mITT) Population consisted of all randomized participants who received study intervention. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 393 | 389
Percentage of participants | 67 | 71
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.0456, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.96 to 1.82] — Analysis performed using logistic regression adjusted for treatment, and both clinical status at Baseline and age group as randomized. Missing data was imputed with monotone discriminant multiple imputation assuming data is missing at random

2. Primary Outcome: Part 2: Percentage of Participants Alive and Free of Respiratory Failure at Day 28
Description: Participants were alive and free of respiratory failure if they were in category 1, 2, 3 or 4 from the GlaxoSmithKline (GSK) modified version ordinal scale adapted from World Health Organization (WHO) scale 2020. The 8-point scale was as follows: 1) Non-hospitalized, no limitation of activity; 2) Non-hospitalized,limitation of activity; 3) Hospitalized, no oxygen therapy; 4) Hospitalized, low-flow oxygen by mask or nasal prongs; 5) Hospitalized, highflow oxygen (>=15L/min), continuous positive airway pressure (CPAP), bilevel positive airway pressure (BIPAP), non-invasive ventilation; 6) Hospitalized, intubation and mechanical ventilation; 7) Hospitalized, mechanical ventilation plus additional organ support; 8) Death. Higher scale indicates higher intensity of respiratory failure. Percentage values are rounded off.
Time Frame: At Day 28
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 170 | 172
Percentage of participants | 51 | 52
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.8574, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.67 to 1.61] — Analysis performed using logistic regression adjusted for treatment, age, and both clinical status at Baseline and sex as randomized. Missing data was imputed with monotone logistic multiple imputation assuming data is missing at random

3. Secondary Outcome: Part 1: Number of Participants Who Died Due to All Causes at Day 60
Description: Number of participants who died due to all causes at Day 60 are reported.
Time Frame: At Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 386 | 373
Participants | 93 | 84
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.2057, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.61 to 1.22] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Part 2: Number of Participants Who Died Due to All Causes at Day 28
Description: Number of participants who died due to all causes at Day 28 is reported
Time Frame: At Day 28
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 170 | 172
Participants | 70 | 63
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.3061, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.50 to 1.24] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Part 2: Number of Participants Who Died Due to All Causes at Day 60
Description: Number of participants who died due to all causes at Day 60 is reported
Time Frame: At Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 170 | 171
Participants | 76 | 74
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.6665, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.59 to 1.41] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Part 1: Time to Death Due to All Causes up to Day 60
Description: Time to death due to all causes was defined as the time (days) from dosing to death, due to any cause, up to (and including) Day 60. Median and inter-quartile range (first quartile and third quartile) of time to death are presented.
Time Frame: Up to Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 93 | 84
Days | NA [NA to NA] — <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived. | NA [NA to NA] — <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived.
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.1942, Regression, Cox — p-value is from a one-sided test; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.65 to 1.18] — Model adjusted analysis performed using a Cox proportional hazards model adjusted by treatment, clinical status at Baseline as randomized and age group as randomized

7. Secondary Outcome: Part 2: Time to Death Due to All Causes up to Day 60
Description: as for outcome 6
Time Frame: Up to Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 76 | 74
Days | NA [16 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived. | NA [16 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived.
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.5324, Regression, Cox — p-value is generated from a two-sided test; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.65 to 1.24] — Model adjusted analysis performed using a Cox proportional hazards model adjusted by treatment, clinical status at Baseline as randomized, sex as randomized and age

8. Secondary Outcome: Part 1: Percentage of Participants Alive and Free of Respiratory Failure at Day 7
Description: as for outcome 2
Time Frame: At Day 7
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 396 | 393
Percentage of participants | 42 | 44
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.2871, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.80 to 1.49] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Part 1: Percentage of Participants Alive and Free of Respiratory Failure at Day 14
Description: as for outcome 2
Time Frame: At Day 14
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 394 | 391
Percentage of participants | 61 | 63
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.1754, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.85 to 1.58] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Part 1: Percentage of Participants Alive and Free of Respiratory Failure at Day 42
Description: as for outcome 2
Time Frame: At Day 42
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 392 | 385
Percentage of participants | 70 | 74
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.0616, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.93 to 1.79] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Part 1: Percentage of Participants Alive and Free of Respiratory Failure at Day 60
Description: as for outcome 2
Time Frame: At Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 386 | 373
Percentage of participants | 74 | 75
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.1830, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.84 to 1.63] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Part 2: Percentage of Participants Alive and Free of Respiratory Failure at Day 7
Description: as for outcome 2
Time Frame: At Day 7
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 173 | 174
Percentage of participants | 28 | 37
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.0831, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.95 to 2.39] — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Part 2: Percentage of Participants Alive and Free of Respiratory Failure at Day 14
Description: as for outcome 2
Time Frame: At Day 14
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 171 | 174
Percentage of participants | 43 | 49
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.2557, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.83 to 2.00] — [estimate comment as in outcome 2, analysis 1]

14. Secondary Outcome: Part 2: Percentage of Participants Alive and Free of Respiratory Failure at Day 42
Description: as for outcome 2
Time Frame: At Day 42
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 170 | 172
Percentage of participants | 54 | 54
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.8560, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.67 to 1.61] — [estimate comment as in outcome 2, analysis 1]

15. Secondary Outcome: Part 2: Percentage of Participants Alive and Free of Respiratory Failure at Day 60
Description: as for outcome 2
Time Frame: At Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 170 | 171
Percentage of participants | 55 | 56
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.7533, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.69 to 1.66] — [estimate comment as in outcome 2, analysis 1]

16. Secondary Outcome: Part 1: Time to Recovery From Respiratory Failure up to Day 28
Description: Time to recovery from respiratory failure was defined as the time (days) from dosing to last recovery from respiratory failure up to (and including) Day 28. Participants were in respiratory failure if they were in category 5 or above from the GlaxoSmithKline (GSK) modified ordinal scale adapted from World Health Organization (WHO) scale 2020. The 8-point scale was as follows: 1) Non-hospitalized, no limitation of activity; 2) Non-hospitalized,limitation of activity; 3) Hospitalized, no oxygen therapy; 4) Hospitalized, low-flow oxygen by mask or nasal prongs; 5) Hospitalized, highflow oxygen (>=15L/min), continuous positive airway pressure (CPAP), bilevel positive airway pressure (BIPAP), non-invasive ventilation; 6) Hospitalized, intubation and mechanical ventilation; 7) Hospitalized, mechanical ventilation plus additional organ support; 8) Death. Median and inter-quartile range (first quartile and third quartile) of time to recovery from respiratory failure are presented.
Time Frame: Up to Day 28
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 263 | 281
Days | 10 [5 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 9 [5 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.0959, Regression, Cox — p-value is from a one-sided test; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.95 to 1.32] — [estimate comment as in outcome 6, analysis 1]

17. Secondary Outcome: Part 2: Time to Recovery From Respiratory Failure up to Day 28
Description: as for outcome 16
Time Frame: Up to Day 28
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 90 | 91
Days | 24 [7 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 22 [5 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.4421, Regression, Cox — p-value is generated from a two-sided test; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.84 to 1.50] — [estimate comment as in outcome 7, analysis 1]

18. Secondary Outcome: Part 1: Percentage of Participants Alive and Independent of Supplementary Oxygen at Day 7
Description: Participants were independent of supplementary oxygen if they were in category 1, 2 or 3 from the GlaxoSmithKline (GSK) modified ordinal scale adapted from World Health Organization (WHO) scale 2020. The 8-point scale was as follows: 1) Non-hospitalized, no limitation of activity; 2) Non-hospitalized,limitation of activity; 3) Hospitalized, no oxygen therapy; 4) Hospitalized, low-flow oxygen by mask or nasal prongs; 5) Hospitalized, highflow oxygen (>=15L/min), continuous positive airway pressure (CPAP), bilevel positive airway pressure (BIPAP), non-invasive ventilation; 6) Hospitalized, intubation and mechanical ventilation; 7) Hospitalized, mechanical ventilation plus additional organ support; 8) Death. Percentage values are rounded off.
Time Frame: At Day 7
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 396 | 393
Percentage of participants | 11 | 12
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.2814, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.73 to 1.80] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: Part 1: Percentage of Participants Alive and Independent of Supplementary Oxygen at Day 14
Description: as for outcome 18
Time Frame: At Day 14
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 394 | 391
Percentage of participants | 37 | 37
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.3901, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.77 to 1.42] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Part 1: Percentage of Participants Alive and Independent of Supplementary Oxygen at Day 28
Description: as for outcome 18
Time Frame: At Day 28
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 393 | 389
Percentage of participants | 57 | 57
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.4763, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.75 to 1.36] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Part 1: Percentage of Participants Alive and Independent of Supplementary Oxygen at Day 42
Description: as for outcome 18
Time Frame: At Day 42
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 392 | 385
Percentage of participants | 63 | 66
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.1973, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.84 to 1.56] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Part 1: Percentage of Participants Alive and Independent of Supplementary Oxygen at Day 60
Description: as for outcome 18
Time Frame: At Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 386 | 373
Percentage of participants | 67 | 71
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.1173, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.88 to 1.67] — [estimate comment as in outcome 1, analysis 1]

23. Secondary Outcome: Part 2: Percentage of Participants Alive and Independent of Supplementary Oxygen at Day 7
Description: as for outcome 18
Time Frame: At Day 7
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 173 | 174
Percentage of participants | 3 | 13
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.0037, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 3.98, 95% CI 2-sided [1.57 to 10.13] — [estimate comment as in outcome 2, analysis 1]

24. Secondary Outcome: Part 2: Percentage of Participants Alive and Independent of Supplementary Oxygen at Day 14
Description: as for outcome 18
Time Frame: At Day 14
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 171 | 174
Percentage of participants | 23 | 28
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.3581, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.77 to 2.06] — [estimate comment as in outcome 2, analysis 1]

25. Secondary Outcome: Part 2: Percentage of Participants Alive and Independent of Supplementary Oxygen at Day 28
Description: as for outcome 18
Time Frame: At Day 28
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 170 | 172
Percentage of participants | 39 | 38
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.9621, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.63 to 1.54] — [estimate comment as in outcome 2, analysis 1]

26. Secondary Outcome: Part 2: Percentage of Participants Alive and Independent of Supplementary Oxygen at Day 42
Description: as for outcome 18
Time Frame: At Day 42
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 170 | 172
Percentage of participants | 46 | 41
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.4167, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.54 to 1.29] — [estimate comment as in outcome 2, analysis 1]

27. Secondary Outcome: Part 2: Percentage of Participants Alive and Independent of Supplementary Oxygen at Day 60
Description: as for outcome 18
Time Frame: At Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 170 | 171
Percentage of participants | 51 | 46
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.3408, Regression, Logistic — p-value is generated from a two-sided test; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.53 to 1.25] — [estimate comment as in outcome 2, analysis 1]

28. Secondary Outcome: Part 1: Time to Last Dependence on Supplementary Oxygen
Description: Time to last dependence on supplementary oxygen was defined as the time (days) from dosing to last dependence on supplementary oxygen up to (and including) Day 28. Median and inter-quartile range (first quartile and third quartile) of time to last dependence on supplementary oxygen are presented.
Time Frame: Up to Day 28
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 223 | 221
Days | 22 [11 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 21 [10 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.4250, Regression, Cox — p-value is from a one-sided test; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.85 to 1.23] — [estimate comment as in outcome 6, analysis 1]

29. Secondary Outcome: Part 2: Time to Last Dependence on Supplementary Oxygen
Description: as for outcome 28
Time Frame: Up to Day 28
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 66 | 68
Days | NA [15 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived. | NA [13 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived.
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.4774, Regression, Cox — p-value is generated from a two-sided test; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.81 to 1.59] — [estimate comment as in outcome 7, analysis 1]

30. Secondary Outcome: Part 1: Percentage of Participants Admitted to Intensive Care Unit (ICU) up to Day 28
Description: Participants who were admitted to the ICU up to (and including) Day 28 were evaluated. Percentage values are rounded off.
Time Frame: Up to Day 28
Population: mITT Population (not in ICU at Baseline) comprised of participants in the mITT population who were not in the ICU at Baseline. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 98 | 95
Percentage of participants | 29 | 16
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.0119, Regression, Logistic — p-value is from a one-sided test; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.18 to 0.89] — [estimate comment as in outcome 2, analysis 1]

31. Secondary Outcome: Part 1: Time to Final ICU Discharge
Description: Time to final ICU discharge was defined as the time from dosing to when the participant is discharged from the ICU for the last time up to (and including) Day 28. Median and inter-quartile range (first quartile and third quartile) of time to final ICU discharge is presented.
Time Frame: Up to Day 28
Population: mITT Population admitted to ICU at Baseline comprised of those participants in mITT who were admitted to ICU at Baseline. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 300 | 300
Days | 13 [7 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 15 [7 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.4404, Regression, Cox — p-value is from a one-sided test; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.83 to 1.24] — [estimate comment as in outcome 6, analysis 1]

32. Secondary Outcome: Part 2: Time to Final ICU Discharge
Description: Time to final ICU discharge was defined as the time from dosing to when the participant was discharged from the ICU for the last time up to (and including) Day 28. Median and inter-quartile range (first quartile and third quartile) of time to final ICU discharge is presented.
Time Frame: Up to Day 28
Population: mITT Population admitted to ICU at Baseline. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 38 | 44
Days | NA [12 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived. | NA [7 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived.
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.6253, Regression, Cox — p-value is generated from a two-sided test; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.72 to 1.72] — [estimate comment as in outcome 7, analysis 1]

33. Secondary Outcome: Part 1: Time to First Discharge From Investigator Site up to Day 60
Description: Time to first discharge from investigator site was defined as the time (days) from dosing to when the participant was first discharged from investigator site (IS) up to (and including) Day 60. Median and inter-quartile range (first quartile and third quartile) of time to first discharge from investigator site is presented.
Time Frame: Up to Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 288 | 294
Days | 18 [11 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 18 [10 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.1078, Regression, Cox — p-value is from a one-sided test; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.94 to 1.30] — [estimate comment as in outcome 6, analysis 1]

34. Secondary Outcome: Part 1: Time to First Discharge to Non-hospitalized Residence up to Day 60
Description: Time to first discharge to non-hospitalized residence was defined as the time (days) from dosing to when the participant was discharged to a non-hospitalized residence for the first time up to (and including) Day 60. Median and inter-quartile range (first quartile and third quartile) of time to first discharge to non-hospitalized residence is presented.
Time Frame: Up to Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 269 | 280
Days | 21 [12 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 20 [11 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.
Statistical Analysis 1: Comparison: Part 1: Placebo 1 vs Part 1: Otilimab 90 mg; Test type: Other; p = 0.1140, Regression, Cox — p-value is from a one-sided test; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.94 to 1.31] — [estimate comment as in outcome 6, analysis 1]

35. Secondary Outcome: Part 2: Time to First Discharge From Investigator Site up to Day 60
Description: Time to first discharge from investigator site was defined as the time (days) from dosing to when the participant was first discharged from investigator site up to (and including) Day 60. Median and inter-quartile range (first quartile and third quartile) of time to first discharge from investigator site is presented.
Time Frame: Up to Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 96 | 99
Days | 36 [15 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 37 [15 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.7084, Regression, Cox — p-value is generated from a two-sided test; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.80 to 1.40] — [estimate comment as in outcome 7, analysis 1]

36. Secondary Outcome: Part 2: Time to First Discharge to Non-hospitalized Residence
Description: as for outcome 34
Time Frame: Up to Day 60
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 86 | 90
Days | NA [18 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived. | 53 [15 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.
Statistical Analysis 1: Comparison: Part 2: Placebo 2 vs Part 2: Otilimab 90 mg; Test type: Other; p = 0.4085, Regression, Cox — p-value is generated from a two-sided test; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.84 to 1.52] — [estimate comment as in outcome 7, analysis 1]

37. Secondary Outcome: Part 1: Number of Participants With Serious Adverse Events (SAEs) and Common (>=5%) Non-serious Adverse Events (Non-SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose may result in death or is life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity or is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment or is associated with liver injury and impaired liver function. Number of participants with any SAE and common (>=5%) non-SAEs are presented.
Time Frame: Up to Day 60
Population: Safety population comprised of all participants who received study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg
Number analyzed (Participants) | 396 | 397
Participants
  Non-SAEs | 67 | 91
  SAEs | 147 | 124

38. Secondary Outcome: Part 2: Number of Participants With SAEs and Common (>=5%) Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose may result in death or is life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity or is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment or is associated with liver injury and impaired liver function. Number of participants with any SAE and common (>=5%) non-SAEs are presented.
Time Frame: Up to Day 60
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
Number analyzed (Participants) | 173 | 174
Participants
  Non-SAEs | 57 | 50
  SAEs | 90 | 90

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs, and non-SAEs were collected up to Day 60 in Part 1 and 2 of the study
Description: SAEs and non-serious AEs were reported for the Safety Population which comprised of all participants who received study intervention. All-cause mortality was reported for Enrolled population (all participants who entered the study). Sixteen participants from Enrolled Population (N=1156) did not receive study treatment, hence were not included in Safety Population (N=1140).
Arm/Group | Part 1: Placebo 1 | Part 1: Otilimab 90 mg | Part 2: Placebo 2 | Part 2: Otilimab 90 mg
All-Cause Mortality (participants affected / at risk) | 93/403 | 84/403 | 76/175 | 74/175
Serious Adverse Events (participants affected / at risk) | 147/396 | 124/397 | 90/173 | 90/174
Other Adverse Events (participants affected / at risk) | 97/396 | 115/397 | 57/173 | 51/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo 1 (N=396) | Part 1: Otilimab 90 mg (N=397) | Part 2: Placebo 2 (N=173) | Part 2: Otilimab 90 mg (N=174)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 17 (18) | 8 (8) | 6 (6)
Multiple organ dysfunction syndrome (General disorders) | 15 (15) | 12 (12) | 8 (8) | 6 (6)
Septic shock (Infections and infestations) | 13 (14) | 14 (14) | 5 (5) | 8 (8)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (9) | 9 (9) | 6 (6)
Pneumonia (Infections and infestations) | 9 (9) | 7 (7) | 5 (5) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 10 (11) | 9 (9) | 1 (1) | 6 (6)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 11 (11) | 3 (3) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 12 (12) | 4 (4) | 5 (5)
COVID-19 (Infections and infestations) | 5 (5) | 3 (3) | 9 (9) | 6 (6)
Cardiac arrest (Cardiac disorders) | 4 (4) | 8 (11) | 7 (9) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 7 (7) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 8 (8) | 1 (1) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 6 (6) | 3 (3) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (2) | 4 (4) | 7 (7)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 5 (5) | 5 (5)
Sepsis (Infections and infestations) | 7 (7) | 1 (1) | 2 (2) | 4 (4)
Pneumonia staphylococcal (Infections and infestations) | 6 (6) | 1 (1) | 1 (1) | 4 (4)
Pneumonia pseudomonal (Infections and infestations) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 4 (4) | 0 (0) | 3 (3) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Klebsiella sepsis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Staphylococcal sepsis (Infections and infestations) | 2 (3) | 3 (3) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Shock haemorrhagic (Vascular disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Pneumonia serratia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Acinetobacter infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Device related bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oxygen consumption increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia proteus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tracheobronchitis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acinetobacter sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Citrobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Citrobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fusobacterium infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis fulminant (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Homeless (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercapnic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lactobacillus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mycetoma mycotic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Organic brain syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumopericardium (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary function test decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serratia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo 1 (N=396) | Part 1: Otilimab 90 mg (N=397) | Part 2: Placebo 2 (N=173) | Part 2: Otilimab 90 mg (N=174)
Constipation (Gastrointestinal disorders) | 35 (35) | 39 (42) | 15 (16) | 16 (16)
Pneumonia (Infections and infestations) | 21 (21) | 37 (43) | 12 (12) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 22 (22) | 18 (19) | 10 (10) | 11 (11)
Acute kidney injury (Renal and urinary disorders) | 17 (18) | 15 (16) | 11 (13) | 8 (9)
Hypotension (Vascular disorders) | 13 (17) | 13 (14) | 11 (13) | 9 (11)
Atrial fibrillation (Cardiac disorders) | 15 (15) | 11 (13) | 10 (11) | 7 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (15) | 12 (13) | 4 (5) | 10 (14)
Urinary tract infection (Infections and infestations) | 13 (13) | 12 (13) | 10 (10) | 5 (5)
Hypernatraemia (Metabolism and nutrition disorders) | 9 (9) | 20 (22) | 1 (1) | 3 (4)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 5 (5) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT04376684/Prot_002.pdf
  • Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT04376684/SAP_003.pdf